CLINICAL TRIAL: NCT06472557
Title: Spinocerebellar Ataxia Type 27B Natural History Study (SCA27B-NHS)
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Matthis Synofzik, Principal Investigator, Leading Consultant, University Hospital Tuebingen
Other Study IDs: SCA27B-NHS
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Spinocerebellar Ataxia Type 27B
Keywords: ataxia; SCA27B; FGF14; Natural History Study; Outcome Validation
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Biosample collection including blood (DNA, serum, plasma, RNA, PBMC) and urine; and optional CSF and skin biopsy
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- SCA27B: Participants with genetically confirmed SCA27B (OMIM 620174), i.e. ≥250 uninterrupted GAA repeat expansions in FGF14, will be recruited. Target sample size for the SCA27B cohort is 200 participants.
- SCA27B risk subjects: First-degree relatives at risk for SCA27B, both with known and unknown carrier status, will be included to capture presymptomatic disease stages. Target sample size for the risk cohort is 50 participants
- Unrelated healthy controls: Unrelated healthy controls may undergo the same study procedures as the SCA27B cohort to determine age-related effects on the multimodal outcomes. Target sample size for the control cohort is 50.

SUMMARY:
This international, multi-center, multi-modal, and prospective observational cohort study aims to validate trial outcomes for capturing disease progression in Spinocerebellar Ataxia Type 27B (SCA27B), with combined multi-modal capture of clinical outcome assessments, digital-motor assessments, and molecular biomarkers.

DETAILED DESCRIPTION:
The investigators will perform an international, multi-center, multi-modal, and registry-based standardized prospective Natural History Study (NHS) in Spinocerebellar Ataxia Type 27B (SCA27B), including the presymptomatic phase of the disease (i.e. presymptomatic subjects at risk for SCA27B). Participants will be assessed annually. Clinical data, including clinician-reported outcomes and patient-focused outcomes, will be entered into a clinical database customized to the requirements of this specific study (SCA27B Registry; www.ataxia-registries.org). Digital-motor outcomes comprise digital gait assessment by wearable sensors, and digital assessment of upper limb movements by Q-Motor. At all study visits, participants will be asked to donate biosamples; and participants can elect to participate in sampling of blood, urine, CSF, and/or a skin biopsy. Based on this multimodal protocol, the study aims to determine the most sensitive, comprehensive, and reliable outcome measures for future therapeutic trials in SCA27B.

ELIGIBILITY:
Inclusion Criteria:

* SCA27B: genetic diagnosis of ≥250 uninterrupted GAA repeat expansions in FGF14
* SCA27B risk subject: asymptomatic first-degree relative of SCA27B participant with known or unknown carrier status
* Unrelated healthy controls: no signs or history of neurological or psychiatric disease AND
* Written informed consent AND
* Participants are willing and able to comply with study procedures

Exclusion Criteria:

* SCA27B: Missing informed consent
* SCA27B risk subjects: Missing informed consent
* Unrelated healthy controls: Missing informed consent, or concurrent neurological, orthopedic, or other diseases interfering with the motor assessments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls participants with clinically manifest and genetically confirmed SCA27B and first-disease relatives at-risk for SCA27B, as well as healthy unrelated controls to contrast unspecific, age- or sex-related findings to disease-related specific findings.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Friedreich Ataxia Rating Scale - Neurological Examination Part E (upright stability) from baseline to 2-year follow-up | 24 months
  Severity of ataxia in the gait and balance domain will be assessed by application of part E of the neurological examination of Friedreich Ataxia Rating Scale (FARS-E). The total score is calculated as the sum of 7 items, yielding a total score between 0 and 28. Hereby, higher FARS-E scores indicate more severe functional impairment.

SECONDARY OUTCOMES:
Change of Scale for the Assessment and Rating of Ataxia (SARA) from baseline to 2-year follow-up | 24 months
  Severity of ataxia will be assessed by application of the Scale for the Assessment and Rating of Ataxia (SARA). The total score is calculated as the sum of 8 items, yielding a total score between 0 and 40. Hereby, higher SARA scores indicate more severe disease.
Friedreich Ataxia Rating Scale - Activities of Daily Living (FARS-ADL) from baseline to 2-year follow-up | 24 months
  Impairment in activities of daily living will be assessed by application of the Activities of Daily Living part of the Friedreich Ataxia Rating Scale (FARS-ADL). The total score is calculated as the sum of 9 items, yielding a total score between 0 and 36. Hereby, higher FARS-ADL scores indicate more severe functional impairment.
Patient Global Impression of Change (PGI-C) from baseline to 1-year and 2-year follow-up | 24 months
  Patient-experienced longitudinal change of ataxia severity will be assessed by asking for the Patient Global Impression of Change (PGI-C) as patient-reported outcome and anchor for longitudinal validation of other outcomes. The PGI-C consists of 7 levels from 1 = very much worse, to 4 = no change, to 7 = very much improved.
Digital gait and balance assessment from baseline to 2-year follow-up | 24 months
  Gait and balance will be assessed digitally with body-worn sensors (inertial measurement units), which record acceleration or rotational movements during specific gait and balance tasks.

OTHER OUTCOMES:
Activities-specific Balance Confidence Scale (ABC Scale) from baseline to 2-year follow-up | 24 months
  Balance problems experienced by the participant will be assessed by application of the Activities-specific Balance Confidence Scale (ABC Scale) as patient-reported outcome. The total score is calculated as the average of 16 items, yielding a total score between 0 and 100% confidence in balance. Hereby, lower scores on the ABC Scales indicate more severe disease.
Friedreich Ataxia Rating Scale - Functional Staging from baseline to 2-year follow-up | 24 months
  Global severity will be assessed by application of the functional staging of the Friedreich Ataxia Rating Scale. The functional staging ranges from 1 (minimal signs detected by physician) to 6 (confined to wheelchair and total dependency). Hereby, higher functional stages indicate more severe functional impairment.
Digital assessment of upper limb movement from baseline to 2-year follow-up | 24 months
  Motor impairment of the upper and lower limb will be assessed digitally with a quantitative motor examination (Q-Motor) of finger tapping, diadochokinesia and visually guided target reaching.

CONTACTS AND LOCATIONS:
Overall Officials: Matthis Synofzik, Prof. Dr., Principal Investigator — University Hospital Tübingen; Andreas Traschütz, Dr. Dr., Principal Investigator — University Hospital Tübingen
Locations (4):
- Department of Neurology, Motol University Hospital, Second Faculty of Medicine, Charles University, Prague, Czechia
- Germany (2):
  - Center for Neurology & Hertie-Institute for Clinical Brain Research, Dept. for Neurodegenerative Diseases, Tübingen, Baden-Wurttemberg
  - Department of Neurology & Center for Translational Neuro- and Behavioral Sciences, Essen University Hospital, University of Duisburg-Essen, Essen, North Rhine-Westphalia
- Department of Neurology, Donostia University Hospital, BioGipuzkoa Health Research Institute, San Sebastián, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request.